CLINICAL TRIAL: NCT04443335
Title: Comparison of Continuous Feeding and Sequential Feeding on Gut Microbiota and Metabolomics in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qingdao University (Other)
Responsible Party: Principal Investigator, Bo Yao,phD, Clinician of critical care medicine, principal investigator, Qingdao University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QYFYKYLL761311920
Record Dates: First submitted 2020-06-21; First posted 2020-06-23 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Feeding Behavior
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- continuous feeding (Sham Comparator): The total amount of every days' Enteral Nutritional Suspension was fed at constant speed for 24h
  Interventions: Behavioral: continous feeding
- sequential feeding (Experimental): This feeding mode utilizes a combination of continuous feeding in the beginning, time-restricted feeding in the second stage and oral feeding in the last stage
  Interventions: Behavioral: sequential feeding

INTERVENTIONS:
Behavioral: continous feeding — At the beginning, all the patients received continuous feeding. After achieving ≥80% of the nutrition target calories (25-30 kcal/kg/d) through continuous feeding, the patients were randomly assigned into the sequential feeding (SF) group or the continuous feeding (CF) group with a random number table. Patients in the CF group received continuous feeding with constant velocity by enteral feeding pump over one day.
  Arms: continuous feeding
Behavioral: sequential feeding — At the beginning, all the patients received continuous feeding. After achieving ≥80% of the nutrition target calories (25-30 kcal/kg/d) through continuous feeding, the patients were randomly assigned into the sequential feeding (SF) group or the continuous feeding (CF) group with a random number table. In the SF group, continuous feeding was changed into time-restricted feeding. The total daily dosage of enteral nutrition was equally distributed during three time periods at 7-9:00, 11-13:00 and 17-19:00. Other times of the day were fasting times. Enteral nutritional suspension in each time period was administered at a uniform rate within two hours by an enteral feeding pump.
  Arms: sequential feeding

SUMMARY:
Continuous feeding is the most popular enteral feeding mode in the ICU because of its lower nursing burden and theoretically better intestinal toleration. However, continuous feeding is nonphysiological. We proposed a feeding mode called sequential feeding, as it utilizes a combination of continuous feeding in the beginning, time-restricted feeding in the second stage, and oral feeding at last.

The gut microbiota plays a critical role in human health due to its many useful functions. Not only dietary structure but also eating mode (eating time for example) influenced the gut microbiota in a healthy population. Therefore, we think this new feeding mode, sequential feeding, also has different influences on gut microbiota and metabolomics in critically ill patients compared to continuous feeding.

DETAILED DESCRIPTION:
Nutrition is an important part of therapy for critically ill patients. Continuous feeding is the most popular enteral feeding mode in the ICU because of its lower nursing burden and theoretically better intestinal toleration. However, continuous feeding is nonphysiological. In our opinion, feeding mode should be changed according to gastrointestinal function and disease progression; one singe feeding mode is not always suitable for critically ill patients. We proposed a feeding mode called sequential feeding, as it utilizes a combination of continuous feeding in the beginning, time-restricted feeding in the second stage, and oral feeding at last.

The gut microbiota plays a critical role in human health due to its many useful functions, such as metabolism, vitamin metabolism, and maintenance of the intestinal barrier and immune system. Not only dietary structure but also eating mode (eating time for example) influenced the gut microbiota in a healthy population. Therefore, we think this new feeding mode, sequential feeding, also has different influences on gut microbiota and metabolomics in critically ill patients compared to continuous feeding.

ELIGIBILITY:
Inclusion Criteria:

●Patients newly admitted to the ICU and fed through gastric tubes

Exclusion Criteria:

* Patients with the ability to eat orally at admission
* Patients with diabetes or gastrointestinal disease
* Patients who are unable to tolerate enteral feeding
* An estimated feeding time of less than 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Shannon index | at the time point of 7th feeding day after achieving ≥80% of the nutrition target calories
  Shannon index is a paramater of α diversity in gut microbiota Full-length 16S rRNA gene sequencing analysis using QIIME software

SECONDARY OUTCOMES:
bacteria bundance | at the time point of 7th feeding day after achieving ≥80% of the nutrition target calories
  It is a paramater of amount of bactera by Full-length 16S rRNA gene sequencing analysis using QIIME software
numbers of compounds | at the time point of 7th feeding day after achieving ≥80% of the nutrition target calories
  it is a paramater by untargeted metabolomics analysis

CONTACTS AND LOCATIONS:
Overall Officials: Bo Yao, phD, Principal Investigator — The affiliated hospital of Qingdao
Locations (1):
- The affiliated hospital of qingdao university, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
connect to corresponding author by email after paper publication
Supporting Information: Study Protocol, CSR
Time Frame: connect to corresponding author by email after paper publication
Access Criteria: by appropriate reasons

REFERENCES:
- [Result] McClave SA, Taylor BE, Martindale RG, Warren MM, Johnson DR, Braunschweig C, McCarthy MS, Davanos E, Rice TW, Cresci GA, Gervasio JM, Sacks GS, Roberts PR, Compher C; Society of Critical Care Medicine; American Society for Parenteral and Enteral Nutrition. Guidelines for the Provision and Assessment of Nutrition Support Therapy in the Adult Critically Ill Patient: Society of Critical Care Medicine (SCCM) and American Society for Parenteral and Enteral Nutrition (A.S.P.E.N.). JPEN J Parenter Enteral Nutr. 2016 Feb;40(2):159-211. doi: 10.1177/0148607115621863. No abstract available. PMID 26773077
- [Result] Singer P, Blaser AR, Berger MM, Alhazzani W, Calder PC, Casaer MP, Hiesmayr M, Mayer K, Montejo JC, Pichard C, Preiser JC, van Zanten ARH, Oczkowski S, Szczeklik W, Bischoff SC. ESPEN guideline on clinical nutrition in the intensive care unit. Clin Nutr. 2019 Feb;38(1):48-79. doi: 10.1016/j.clnu.2018.08.037. Epub 2018 Sep 29. PMID 30348463
- [Result] Lynch SV, Pedersen O. The Human Intestinal Microbiome in Health and Disease. N Engl J Med. 2016 Dec 15;375(24):2369-2379. doi: 10.1056/NEJMra1600266. No abstract available. PMID 27974040
- [Result] McDonald D, Ackermann G, Khailova L, Baird C, Heyland D, Kozar R, Lemieux M, Derenski K, King J, Vis-Kampen C, Knight R, Wischmeyer PE. Extreme Dysbiosis of the Microbiome in Critical Illness. mSphere. 2016 Aug 31;1(4):e00199-16. doi: 10.1128/mSphere.00199-16. eCollection 2016 Jul-Aug. PMID 27602409
- [Result] Kaczmarek JL, Thompson SV, Holscher HD. Complex interactions of circadian rhythms, eating behaviors, and the gastrointestinal microbiota and their potential impact on health. Nutr Rev. 2017 Sep 1;75(9):673-682. doi: 10.1093/nutrit/nux036. PMID 28938796
- [Derived] Yao B, Liu JY, Liu Y, Song XX, Wang SB, Liu N, Dong ZH, Yuan ZY, Han XN, Xing JY. Sequential versus continuous feeding and its effect on the gut microbiota in critically ill patients: A randomized controlled trial. Clin Nutr ESPEN. 2025 Apr;66:245-254. doi: 10.1016/j.clnesp.2025.01.019. Epub 2025 Jan 9. PMID 39798866